CLINICAL TRIAL: NCT05761561
Title: Trial of Exercise and Lifestyle (TEAL) for Women With Ovarian and Endometrial Cancer
Brief Title: Trial of Exercise and Lifestyle for Women With Ovarian and Endometrial Cancer
Acronym: TEAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of Miami (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20211179; U01CA271278 (NIH)
Record Dates: First submitted 2023-02-06; First posted 2023-03-09 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and medical nutrition (Experimental): Over the intervention period (18 weeks on average - dependent on length of chemotherapy) women in the intervention arm will receive weekly counseling sessions, the study dietitian and exercise trainer will each conduct weekly sessions to assist the participants in achieving the diet and exercise study goals.
  Interventions: Behavioral: Exercise and medical nutrition
- Control (No Intervention): Contact limited to study assessments.

INTERVENTIONS:
Behavioral: Exercise and medical nutrition — The study dietitian and exercise trainer will each conduct weekly counseling sessions via telephone or zoom throughout the course of chemotherapy (approximately 18 weeks) to assist the participants in achieving the diet and exercise study goals. Participants will be provided written informational material, exercise bands for strength training and a Fitbit to record activity.
  Participant goals are to: 1) participate in 150 min/week of moderate-intensity physical activity 2) participate in two weekly strength training sessions; 3) eat a combination of 5 or more servings of vegetables and/or fruits per day 4) consume 25 grams or more of fiber/day; 5) consume adequate amounts of protein to prevent muscle wasting (1.2g/kg body weight).
  Arms: Exercise and medical nutrition

SUMMARY:
An anticipated 200 women with newly diagnosed ovarian and endometrial cancer scheduled to receive chemotherapy (adjuvant chemotherapy after surgery or neoadjuvant chemotherapy before surgery) will be recruited from Smilow Cancer Hospital Network at Yale Cancer Center (YCC) and Sylvester Comprehensive Cancer Center (SCCC) at University of Miami.

Participants will be randomized to an exercise and medical nutrition intervention arm with weekly counseling sessions throughout chemotherapy, or a control arm.

Study assessments will be conducted at baseline, post-chemotherapy/end of intervention and at 1-year post diagnosis. Women who are prescribed neoadjuvant therapy will have additional assessments prior to surgery.

Data required to calculate the primary endpoint (relative dose intensity of chemotherapy) will be abstracted from the medical record directly following each chemotherapy session.

DETAILED DESCRIPTION:
200 women with newly diagnosed ovarian or endometrial cancer scheduled to receive chemotherapy (adjuvant chemotherapy after surgery or neoadjuvant chemotherapy before surgery) will be recruited from Smilow Cancer Hospital at Yale Cancer Center (YCC) and Sylvester Comprehensive Cancer Center (SCCC) at University of Miami. If women are interested and eligible, the study team will obtain consent and collect baseline data. Participants will be randomized to an exercise and medical nutrition intervention (18 weeks dependent on length of chemotherapy) or usual care throughout therapy. After the standard 6 cycles of chemotherapy (~18 weeks), a post-chemotherapy/end of intervention visit will be conducted. Follow-up assessments will be at standard of care visits (12-months post-diagnosis). Data required to calculate the primary endpoint (relative dose intensity of chemotherapy) will be abstracted from the medical record directly following each chemotherapy session.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of epithelial ovarian cancer, fallopian tube or primary peritoneal carcinoma, stage I-IV OR have a diagnosis of advanced or metastatic endometrial carcinoma (including carcinosarcoma) AND their treatment regimen includes carboplatin and taxane (or equivalent)
* be scheduled to receive at least 6 cycles of neoadjuvant or adjuvant chemotherapy
* be physically able to walk without a walking aid (e.g. cane or walker)
* be able to complete forms, understand instructions and read intervention book in English or Spanish
* agree to be randomly assigned to either group
* have clearance from oncologist to participate
* be ≥ 18 years of age

Exclusion Criteria:

* having already completed a 2nd cycle of chemotherapy
* already practicing dietary (>7 servings of fruits and vegetables per day) OR physical activity guidelines (≥150 min per week of moderate to vigorous exercise and resistance training two times per week) since diagnosis
* pregnancy or intention to become pregnant
* recent (past year) stroke/myocardial infarction or congestive heart failure/ejection fraction <40%
* presence of dementia or major psychiatric disease
* in active treatment including target or biologic therapies for any other cancer (excluding hormone therapy treatments)
* receiving external beam radiation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy completion rate (relative dose intensity) | Through end of first line chemotherapy, an average of 5 months
  Chemotherapy completion rate will be assessed as the average relative dose intensity for the originally planned regimen based on standard formulas. This will be measured using the number and percent of patients requiring dose-adjustments, dose-delays, reason for dose.

SECONDARY OUTCOMES:
Change in Skeletal muscle mass | Through study completion, an average of 1 year
  Skeletal muscle mass will be assessed assessed using CT scans. The L3 slice used for analysis will be within 3-5mm of the lower border of the L3 vertebral body across individuals. A multiple-step procedure will be used to segment images into skeletal muscle, excluding visceral adipose tissue, subcutaneous adipose tissue, organs, vessels, and bony structures.
Change in Muscle Mass assessed using D3Creatine dilution method | Through end of first line chemotherapy, an average of 5 months.
  A capsule of D3Creatine will be given to the participant to ingest. Fasting urine sample is then collected between 2-5 days after the dose is ingested and sent for analysis. For subsequent measurements, there is some residual D3Cr remaining in muscle, so a pre- D3Creatine dose urine sample is needed to measure the D3Cr enrichment from the initial dose and a sample taken 2-5 days after the dose.
Change in Healthy Eating Index-2020 (24-hour recall) | Through study completion, an average of 1 year
  24-Hour Dietary Recall will be assessed. Two 24-hour recalls (1 weekday and weekend day, 30-40 minutes to complete) will be captured. Interviewers record all food and beverage consumption over a 24-hour period using the USDA multi-pass method with the University of Minnesota Nutrition Data System-Research Version system. The two days at each time point will be averaged and calories (kcal), nutrients, and diet quality assessed. Diet quality will be calculated using the HEI-2020; range of 0 - 100, higher score indicating better diet quality.
Change in Healthy Eating Index-2020 (FFQ) | Through study completion, an average of 1 year
  Recent diet will be assessed via food frequency questionnaire (FFQ). Diet quality will be calculated using the HEI-2020; range of 0 - 100, higher score indicating better diet quality.
Change in Physical activity - objective measure | Through study completion, an average of 1 year
  Participants will receive an Actigraph GTX9 accelerometer and instructed to wear it on the waist for 7 continuous days. From the Actigraph GTX9, daily summary moderate to vigorous physical activity will be calculated.
Change in Physical activity - subjective measure | Through study completion, an average of 1 year
  Physical Activity Recall: The interviewer administered modified physical activity questionnaire (MPAQ) will measure physical activity.
Change in Neuropathy | Through study completion, an average of 1 year
  The Functional Assessment of Cancer Therapy (FACT)-neuropathy subscale (FACT-GOG-Ntx) will be used to assess neuropathy (38 items).
Change in Cognitive function | Through study completion, an average of 1 year
  Cognitive function will be assessed using the Functional Assessment of Cancer Therapy (FACT)-Cog. This self-administered questionnaire includes four subscales, 'Perceived Cognitive Impairments' (20 items), 'Impact of Quality of Life' (4 items) , 'Comments from Others' (4 items), and 'Perceived Cognitive Abilities' (9 items).
Change in Arthralgia | Through study completion, an average of 1 year
  Arthralgia: Arthralgia will be assessed via the Brief Pain Inventory.
Change in GI disturbance | Through study completion, an average of 1 year
  The 13-item Gastrointestinal Symptom Rating Scale developed for patients with Irritable Bowel Syndrome (GSRS-IBS)with subscales on satiety, abdominal pain, diarrhea, constipation, and bloating, will be used to assess GI disturbance.
Change in lower leg lymphedema | Through study completion, an average of 1 year
  Lower leg lymphedema will be assessed using Gynecology Oncology Cancer Lymphedema Questionnaire.
Change in BMI | Through study completion, an average of 1 year
  Participants will be weighed in light clothing, without shoes, rounding up to the nearest 0.1 kg. Height will be measured without shoes, using a stadiometer, rounding up to the nearest 0.1 cm. BMI will be calculated from the measured weight and height.
Change in waist circumference | Through study completion, an average of 1 year
  Waist measurement will rounded up to the nearest millimeter.
Change in Skin Carotenoids | Through study completion, an average of 1 year
  The Veggie meter will be used to measure carotenoid levels. This method is rapid and non-invasive, and measures skin carotenoids using optical signals.
Change in Fitness | Through study completion, an average of 1 year
  Participants will be complete a 6-minute walk test following the American Thoracic Society's standardized protocol, with the score equal to the distance walked in 6 minutes in meters.
Change in grip strength | Through study completion, an average of 1 year
  Grip strength assessed by dynamometer. Handgrip strength is a valid, simple measure of muscle strength that correlates well with leg strength, poor mobility, and incident disability in activities of daily living.
Change in blood biomarkers | Through study completion, an average of 1 year
  Bloods will be taken. Plasma, serum and buffy coat samples will be prepared and frozen at -80 degrees C. Potential blood biomarkers include: glucose, insulin, leptin, VEGF, CRP, IL-6, TNF-α, CA-125.
Change in financial toxicity | Through study completion, an average of 1 year
  Financial toxicity will be assessed using the Functional Assessment of Chronic Illness Therapy-COST (FACIT-COST), a measure of financial toxicity (financial distress). Values : minimum = 0 and maximum = 48. Higher scores are worse outcome.
Change in level of function and ability to perform specific tasks | Through study completion, an average of 1 year
  Women will complete the Functional Assessment of Cancer Therapy (FACT)-ovarian cancer subscale (FACT-O) (ovarian cancer patients) or the FACT-endometrial (FACT-EN) cancer subscale (endometrial cancer patients) to assess level of function and ability to perform specific tasks.
Change in Social Support | Through study completion, an average of 1 year
  Women will complete the MOS Social Support Survey Subscale.
Change in Social Activity | Through study completion, an average of 1 year
  Women will complete the MOS Social Activity limitations Scale.
Change in Quality of life (SF-36) | Through study completion, an average of 1 year
  Women will complete the Short Form Survey (SF-36) (36 items)
Change in Sleep Quality | Through study completion, an average of 1 year
  Sleep Quality: Women will complete Pittsburgh Sleep Quality Index (PSQI).
Change in Fatigue | Through study completion, an average of 1 year
  Fatigue: Women will complete Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue). Values : minimum = 0 and maximum = 52. Higher scores are worse outcome.
Change in symptoms of chemotherapy assessed using the Common Terminology Criteria for Adverse Events (CTCAE) | Through end of chemotherapy, an average of 5 months.
  The Common Terminology Criteria for Adverse Events (CTCAE) will be used to assess symptoms. This well-validated survey includes symptoms and adverse events related to chemotherapy. The constructs we will measure include dry mouth, mouth/throat sores, taste, appetite, nausea, vomiting, heartburn, constipation, diarrhea, abdominal pain, shortness of breath, dizziness, neuropathy, concentration, memory, pain, insomnia, anxiety, hot flashes and fatigue.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: Undecided
Before making the data available to researchers not involved in the proposed study, we will ensure that the data to be shared are de-identified and comply with both IRB regulations and the Privacy Rule under HIPAA regulations. Under no circumstances will personal identifying information, such as name, address, telephone, medical record number be shared with anyone outside our research team.